CLINICAL TRIAL: NCT01636687
Title: A Randomized, Double-blind, Placebo Controlled, Multicenter Study of Subcutaneous Secukinumab in Autoinjectors to Demonstrate Efficacy After Twelve Weeks of Treatment, and to Assess the Safety, Tolerability, Usability and Long-term Efficacy in Subjects With Chronic Plaque-type Psoriasis
Brief Title: Judging the Efficacy of Secukinumab in Patients With Psoriasis Using AutoiNjector: a Clinical Trial Evaluating Treatment Results (JUNCTURE)
Acronym: JUNCTURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457A2309; 2012-002609-22 (EudraCT Number)
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Plaque-type Psoriasis
Keywords: Psoriasis; Moderate to Severe Plaque-type Psoriasis; Skin condition; skin disease; itching condition; psoriasis vulgaris; relapsing/remitting psoriasis; immune-mediated systemic disease; skin lesions; red skin lesions; scaly patches; papules; plaques; itching
MeSH Terms: conditions — Psoriasis; Skin Diseases; Recurrence; Plaque, Amyloid; Pruritus | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects who were in placebo at Week 52 cannot continue in the extension treatment period
  Interventions: Drug: Placebo
- Secukinumab 150 mg (Experimental): After the data base lock of week 52 data has been performed, subjects received secukinumab 150 mg treatment as open label for the remainder of the extension treatment period.
  Interventions: Drug: Secukinumab 150mg
- Secukinumab 300 mg (Experimental): After the data base lock of week 52 data has been performed, subjects received secukinumab 300 mg treatment as open label for the remainder of the extension treatment period.
  Interventions: Drug: Secukinumab 300mg

INTERVENTIONS:
Drug: Placebo — 2 injections of placebo to secukinumab 150mg per dose
  Arms: Placebo
Drug: Secukinumab 150mg — Secukinumab 150mg: 1 injection of 150 mg secukinumab and 1 injection of placebo to secukinumab 150mg per dose. After Week 52 database lock, study is open label so only 1 injection of secukinumab 150mg per dose were administered
  Arms: Secukinumab 150 mg
Drug: Secukinumab 300mg — Secukinumab 300mg (2 injections of 150mg secukinumab per dose)
  Arms: Secukinumab 300 mg

SUMMARY:
The purpose of this study was to demonstrate efficacy of autoinjector administered secukinumab at Week 12 based on PASI and IGA response rates versus placebo in subjects with moderate to severe chronic plaque-type psoriasis.

ELIGIBILITY:
Inclusion criteria:

* Moderate and severe plaque-type psoriasis diagnosed for at least 6 months.
* Severity of psoriasis disease meeting all of the following three criteria:

  * Psoriasis Area and Severity Index (PASI) score of 12 or greater
  * Investigator's Global Assessment (IGA) score of 3 or greater
  * Total body surface area (BSA) affected of 10% or greater
* Inadequate control by prior use of topical treatment, phototherapy and/or systemic therapy.

Exclusion criteria:

* Current forms of psoriasis other than chronic plaque-type psoriasis (for example, pustular, erythrodermic, guttate).
* Current drug-induced psoriasis.
* Previous use of secukinumab or any drug that targets IL-17 or IL-17 receptor.
* Significant medical problems such as uncontrolled hypertension, congestive heart failure or a condition that significantly immunocompromises the subject.
* Hematological abnormalities.
* History of an ongoing, chronic or recurrent infectious disease, or evidence of untreated tuberculosis.
* History of lymphoproliferative disease or history of malignancy of any organ system within the past 5 years.
* Pregnant or nursing (lactating) women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2012-10-17 (Actual); Primary Completion 2016-10-27 (Actual); Study Completion 2016-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- United States (11):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Johnston, Rhode Island
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Norfolk, Virginia
- Canada (6):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Mississauga, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Novartis Investigative Site, Tallinn, Estonia
- France (3):
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Toulouse
- Germany (14):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Selters
  - Novartis Investigative Site, Tübingen

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Sticherling M, Nikkels AF, Hamza AM, Kwong P, Szepietowski JC, El Sayed M, Ghislain PD, Khotko AA, Patekar M, Ortmann CE, Forrer P, Papanastasiou P, Keefe D. Secukinumab in Pediatric Patients with Plaque Psoriasis: Pooled Safety Analysis from Two Phase 3 Randomized Clinical Trials. Am J Clin Dermatol. 2023 Sep;24(5):821-835. doi: 10.1007/s40257-023-00782-8. Epub 2023 Jun 21. PMID 37341961
- [Derived] Merola JF, McInnes IB, Deodhar AA, Dey AK, Adamstein NH, Quebe-Fehling E, Aassi M, Peine M, Mehta NN. Effect of Secukinumab on Traditional Cardiovascular Risk Factors and Inflammatory Biomarkers: Post Hoc Analyses of Pooled Data Across Three Indications. Rheumatol Ther. 2022 Jun;9(3):935-955. doi: 10.1007/s40744-022-00434-z. Epub 2022 Mar 19. PMID 35305260
- [Derived] Houghton K, Patil D, Gomez B, Feldman SR. Correlation Between Change in Psoriasis Area and Severity Index and Dermatology Life Quality Index in Patients with Psoriasis: Pooled Analysis from Four Phase 3 Clinical Trials of Secukinumab. Dermatol Ther (Heidelb). 2021 Aug;11(4):1373-1384. doi: 10.1007/s13555-021-00564-2. Epub 2021 Jun 10. PMID 34110605
- [Derived] Menter A, Cather JC, Jarratt M, Meng X, Guana A, Nyirady J. Efficacy of Secukinumab on Moderate-to-severe Plaque Psoriasis Affecting Different Body Regions: a Pooled Analysis of Four Phase 3 Studies. Dermatol Ther (Heidelb). 2016 Dec;6(4):639-647. doi: 10.1007/s13555-016-0140-7. Epub 2016 Aug 30. PMID 27576559
- [Derived] Kircik L, Fowler J, Weiss J, Meng X, Guana A, Nyirady J. Efficacy of Secukinumab for Moderate-to-Severe Head and Neck Psoriasis Over 52 Weeks: Pooled Analysis of Four Phase 3 Studies. Dermatol Ther (Heidelb). 2016 Dec;6(4):627-638. doi: 10.1007/s13555-016-0139-0. Epub 2016 Aug 30. PMID 27573260
- [Derived] Paul C, Lacour JP, Tedremets L, Kreutzer K, Jazayeri S, Adams S, Guindon C, You R, Papavassilis C; JUNCTURE study group. Efficacy, safety and usability of secukinumab administration by autoinjector/pen in psoriasis: a randomized, controlled trial (JUNCTURE). J Eur Acad Dermatol Venereol. 2015 Jun;29(6):1082-90. doi: 10.1111/jdv.12751. Epub 2014 Sep 22. PMID 25243910

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 59 placebo subjects completed induction phase. These 59 entered maintenance phase. Of those, 28 were assigned to 150mg AIN457 and 28 were assigned to 300 mg AIN457, while 3 remained with PLC treatment.
Pre-assignment Details: A total of 220 patients were screened at 39 study centers, and 182 patients were randomized at 38 study centers to 3 balanced groups.
Groups:
- AIN457 150 mg: Patients received one secukinumab 150 mg s.c. injection plus one placebo secukinumab s.c. injection at each dosing. In the open label phase only one 150 mg s.c. injection at each dosing.
- AIN457 300 mg: Patients received two secukinumab 150 mg s.c. injections at each dosing. In the open label phase only two 150 mg s.c. injections at each dosing.
- Placebo - AIN457 150 mg: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12, were re randomized to AIN457 150 mg for the remainder of the study.
- Placebo - AIN457 300mg: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12, were re randomized to AIN457 300 mg for the remainder of the study.
- Placebo: placebo secukinumab (2 s.c. injections) at each dosing
Period: Induction Period
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg | Placebo
Started | 61 | 60 | 0 | 0 | 61
Completed | 58 | 60 | 0 | 0 | 59
Not Completed | 3 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg | Placebo
Started | 58 | 60 | 28 | 28 | 3
Completed | 50 | 58 | 26 | 28 | 1
Not Completed | 8 | 2 | 2 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Period: Extension Period
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg | Placebo
Started | 47 | 54 | 25 | 28 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 47 | 54 | 25 | 28 | 0
Not completed — technical problems | 0 | 1 | 2 | 1 | 0
Not completed — Adverse Event | 4 | 3 | 2 | 1 | 0
Not completed — Lack of Efficacy | 7 | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0
Not completed — study terminated by sponsor | 33 | 50 | 17 | 23 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0
Period: Follow-up Period
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg | Placebo
Started | 38 | 45 | 21 | 20 | 2
Completed | 37 | 45 | 21 | 20 | 1
Not Completed | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized set for on treatment groups
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | Total
Number analyzed (Participants) | 61 | 60 | 61 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (14.41) | 46.6 (14.23) | 43.7 (12.74) | 44.7 (13.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 14 | 23 | 57
  Male | 41 | 46 | 38 | 125

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area and Severity Index (PASI) 75 Response and Investigators' Global Assessment (IGA) Mod 2011 0 or 1 Response
Description: Efficacy of secukinumab compared to placebo in subjects with moderate to severe chronic plaque-type psoriasis.
  PASI score was based on assessment of the head, trunk, upper limbs and lower limbs for erythema, thickening (plaque elevation, induration), and scaling (desquamation). PASI scores can range from 0, corresponding to no signs of psoriasis, up to a theoretical maximum of 72.0. PASI-based secondary variables included absolute PASI score, response rates for PASI 75. PASI 50 and PASI 90 were defined as ≥ 50% and ≥ 90% improvement from Baseline in PASI score, respectively, while PASI 100 response corresponded to complete clearing of psoriasis (PASI = 0). IGA mod 2011 was used to evaluate the overall severity of psoriatic disease, with scores ranging from 0 (clear) to 4 (severe). Treatment success was defined as achievement of IGA mod 2011 0 or 1 score.
Time Frame: 12 weeks
Population: Full Analysis Set (FAS) comprises of all patients to whom study treatment has been assigned.
Measure: Number; unit: Percentages of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 60 | 60 | 61
Percentages of participants
  PASI 75 | 71.7 | 86.7 | 3.3
  IGA 0/1 | 53.3 | 73.3 | 0.0
Statistical Analysis 1: Comparison: AIN457 150 mg vs Placebo; Response criterion: IGA 0/1; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Risk Difference (RD) = 53.3, 95% CI 2-sided [36.6 to 67.7]
Statistical Analysis 2: Comparison: AIN457 300 mg vs Placebo; Response Criterion: IGA 0/1; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Risk Difference (RD) = 73.3, 95% CI 2-sided [58.8 to 83.9]
Statistical Analysis 3: Comparison: AIN457 150 mg vs Placebo; Response criterion: PASI 75; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Risk Difference (RD) = 68.4, 95% CI 2-sided [53.1 to 79.8]
Statistical Analysis 4: Comparison: AIN457 300 mg vs Placebo; Response criterion: PASI 75; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Risk Difference (RD) = 83.4, 95% CI 2-sided [70.7 to 91.7]

2. Secondary Outcome: Percentages of Subjects With Successful Self-administration of Study Drug at Week 1
Description: To assess the subject's ability to follow instructions for use with the secukinumab autoinjector
Time Frame: Week 1
Population: Safety set: The safety set included all patients who took at least one dose of study treatment during the treatment period. Patients were analyzed according to treatment received.
Measure: Number; unit: Percentages of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 61 | 60 | 60
Percentages of participants | 100 | 100 | 100

3. Secondary Outcome: Percentage of Subjects With Possible Use-related Hazards
Description: To assess potential use-related hazards with the secukinumab autoinjector for the subject.
Time Frame: Week 1
Population: Safety set
Measure: Number; unit: Percentages of participants
Units Other Than Participants: Participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 61 | 60 | 61
Number analyzed (Participants) | 59 | 58 | 60
Percentages of participants
  Needle stick in a critical area | 0 | 0 | 0
  Needle stick in non-critical area | 0 | 0 | 0
  Any part of the device swallowed | 0 | 0 | 0
  Allergic reaction to devise material | 0 | 0 | 0
  Pain due to bent needle | 0 | 0 | 0
  Any breakage of the device | 0 | 0 | 0
  Swallowing of material debris observed | 0 | 0 | 0
  Any other problem | 0 | 5.1 | 0
  Less than full dose administered | 0 | 1.7 | 0

4. Secondary Outcome: Absolute Change From Baseline in Self-Injection Assessment Questionnaire (SIAQ) Domain Scores at Week 12
Description: The three domains of the POST SIAQ are feelings about injections, self-image, self-confidence, injection-site reactions, ease of use, and satisfaction with self-injection. The SIAQ items are scored on a semantic Likert-type scale where lower numbers indicate a worse experience. Domain scores range from 0 to 10; "0" corresponds to worst experience while "10" corresponds to best experience. Subjects self-injecting at this visit completed this SIAQ questionnaire. The POST-SIAQ is taken after the injection at that visit.
Time Frame: Week 12
Population: Safety Set
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 61 | 60 | 61
Score
  Feelings about injections: number analyzed (Participants) | 54 | 59 | 58
  Feelings about injections | 0.94 (2.190) | 1.13 (1.796) | 0.93 (1.887)
  Self confidence: number analyzed (Participants) | 54 | 60 | 59
  Self confidence | 1.76 (1.763) | 1.68 (1.901) | 1.00 (2.098)
  Satisfaction with self-injection: number analyzed (Participants) | 53 | 58 | 57
  Satisfaction with self-injection | 2.74 (2.741) | 2.63 (2.361) | 1.71 (2.679)

5. Secondary Outcome: Absolute Change From Baseline in Self-Injection Assessment Questionnaire (SIAQ) Domain Scores at Week 48
Description: as for outcome 4
Time Frame: Absolute change from baseline at week 48
Population: Safety set
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Placebo - AIN457 300 mg: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12, were re randomized to AIN457 150 mg for the remainder of the study.
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg | Placebo
Number analyzed (Participants) | 58 | 60 | 28 | 28 | 3
Score
  Feelings about injections | 0.92 (1.853) | 1.34 (2.336) | 1.43 (2.049) | 0.73 (1.450) | 0.42 (1.768)
  Self confidence | 1.88 (1.926) | 1.86 (2.052) | 1.17 (3.033) | 1.70 (2.145) | 0.00 (3.536)
  Satisfaction with self-injection | 2.93 (2.853) | 2.50 (2.121) | 2.29 (2.650) | 1.98 (2.853) | 2.50 (0.000)

6. Secondary Outcome: Percentages of Participants With PASI 50, PASI 75, PASI 90, PASI 100 and IGA Mod 2011 0 or 1 Response - Induction Period
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 50, 75, 90 and 100 were defined as participants achieving ≥ 50%, 75%, 90% or 100% improvement from baseline.
  The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe.
Time Frame: Week 12
Population: Full Analysis Set (FAS)
Measure: Number; unit: Percentages of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 61 | 60 | 61
Percentages of participants
  PASI 50 | 78.3 | 96.7 | 8.2
  PASI 90 | 40.0 | 55.0 | 0.0
  PASI 100 | 16.7 | 26.7 | 0.0

7. Secondary Outcome: Percentages of Participants With PASI 50, PASI 75, PASI 90, PASI 100 and IGA Mod 2011 0 or 1 Response - Maintenance Period (Observed Data)
Description: as for outcome 6
Time Frame: Week 12 up to Week 52
Population: Full Analysis Set (FAS). Results after Week 160 and beyond cannot be interpreted meaningfully due to low number of evaluable patients at these visits.
Measure: Number; unit: Percentages of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 61 | 60 | 28 | 28
Percentages of participants
  Week 52 IGA 0/1 | 64.7 | 70.7 | 56.0 | 85.7
  Week 52 PASI 75 | 82.4 | 82.8 | 76.0 | 96.4
  Week 52 PASI 50 | 96.1 | 94.8 | 88.0 | 100.0
  Week 52 PASI 90 | 62.7 | 65.5 | 52.0 | 89.3
  Week 52 PASI 100 | 35.3 | 39.7 | 40.0 | 64.3

8. Secondary Outcome: Absolute Change From Baseline for PASI Score - Induction Period
Description: PASI: Combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section(head:01, arms:0.2 body:0.3 legs:0.4)
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 61 | 60 | 61
Units on a scale | -15.52 (7.841) | -16.67 (6.552) | -1.26 (6.621)

9. Secondary Outcome: Absolute Change From Baseline for PASI Score Over Time up to Week 52 - Maintenance Period (Observed Data)
Description: Psoriasis Area and Severity Index (PASI): Combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section(head:01, arms:0.2 body:0.3 legs:0.4).
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg
Number analyzed (Participants) | 61 | 60 | 28 | 28
Units on a scale | -18.3 (6.75) | -16.4 (5.99) | -15.2 (5.85) | -18.8 (5.59)

10. Secondary Outcome: Percentage of Participants in Each IGA Mod 2011 Category - Induction Period
Description: The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe
Time Frame: Week 12
Population: Full Analysis Set (FAS) - All patients to whom study treatment was assigned.
Measure: Number; unit: Percentages of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 61 | 60 | 61
Percentages of participants
  clear: number analyzed (Participants) | 60 | 60 | 61
  clear | 18.3 | 30.0 | 0.0
  almost clear: number analyzed (Participants) | 60 | 60 | 61
  almost clear | 35.0 | 45.0 | 0.0
  mild: number analyzed (Participants) | 60 | 60 | 61
  mild | 25.0 | 18.3 | 8.2
  moderate: number analyzed (Participants) | 60 | 60 | 61
  moderate | 15.0 | 6.7 | 60.7
  severe: number analyzed (Participants) | 60 | 60 | 61
  severe | 6.7 | 0.0 | 31.1

11. Secondary Outcome: Percentages of Participants in Each IGA Mod 2011 Category Over Time up to Week 52 - Maintenance Period (Observed Data)
Description: The Investigators' Global Assessment (IGA) mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe.
Time Frame: Week 52
Population: Full Analysis Set (FAS)
Measure: Number; unit: Percentages of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg
Number analyzed (Participants) | 61 | 60 | 28 | 28
Percentages of participants
  Clear | 35.3 | 39.7 | 40.0 | 64.3
  Almost clear | 29.4 | 31.0 | 16.0 | 21.4
  Mild | 19.6 | 19.0 | 24.0 | 10.7
  Moderate | 11.8 | 6.9 | 20.0 | 3.6
  Severe | 3.9 | 3.4 | 0.0 | 0.0

12. Secondary Outcome: Change From Baseline in EQ-5D up to Week 12 - Induction Period
Description: ED-5Q: Participant rated questionnaire to assess health related quality of life in terms of a single utility score. Five domains are assessed mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each with three possible score: 1 indicates no problems, better state of health; 3 indicates worst state of health (example "confined to bed") A visual analog scale (VAS) assesses the health status from 0 (worst possible health state) to 100 (best possible health state).
Time Frame: Week 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 61 | 60 | 61
unit on a scale | 13.5 (19.63) | 15.3 (19.80) | -0.5 (14.89)

13. Secondary Outcome: Change From Baseline in EQ-5D Over Time up to Week 52 - Maintenance Period
Description: as for outcome 12
Time Frame: Week 52
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg | Placebo
Number analyzed (Participants) | 61 | 60 | 28 | 28 | 3
unit on a scale | 16.8 (20.34) | 17.4 (20.38) | 12.9 (28.45) | 9.9 (10.94) | 10.0 (9.00)

14. Secondary Outcome: Percentage Changes From Baseline in Dermatology Life Quality Index (DLQI) Score - Induction Period
Description: The DLQI is a quality of life measure used in the psoriatic The 10-item questionnaire has a score range of 0 (best) to 30 (worst) with higher scores indicating poor quality of life. The instrument contains six functional scales (i.e., symptoms and feeling, daily activities, leisure, work and school, personal relationships, treatment). Each item has 4 response categories, ranging from 0 (not at all) to 3 (very much). "Not relevant" is also a valid response and is scored as 0. The DLQI total score is a sum of the 10 questions.
  A negative median percent change from baseline indicates improvement.
Time Frame: Baseline, up to Week 12
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 56 | 55 | 55
percent change | -83.3 [-88.9 to -75.0] | -86.8 [-95.0 to -82.5] | -17.9 [-32.7 to -1.1]

15. Secondary Outcome: Percentage Changes From Baseline in Dermatology Life Quality Index (DLQI) Score Over Time up to Week 52 - Maintenance Period
Description: as for outcome 14
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg | Placebo
Number analyzed (Participants) | 56 | 55 | 25 | 27 | 3
Percent change | -90.9 [-95.0 to -85.0] | -91.2 [-94.7 to -84.2] | -78.5 [-90.0 to -59.5] | -97.7 [-100 to -81.3] | -53.7 [-72.7 to NA] — Too few events to calculate the upper limit.

16. Secondary Outcome: Percentage of Participants Achieving a DLQI Score of 0 or 1 at Week 12 - Induction Period
Description: The DLQI is a quality of life measure used in the psoriatic The 10-item questionnaire has a score range of 0 (best) to 30 (worst) with higher scores indicating poor quality of life. The instrument contains six functional scales (i.e., symptoms and feeling, daily activities, leisure, work and school, personal relationships, treatment). Each item has 4 response categories, ranging from 0 (not at all) to 3 (very much). "Not relevant" is also a valid response and is scored as 0. The DLQI total score is a sum of the 10 questions.
Time Frame: Week 12
Population: Full analysis set (FAS)
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 59 | 59 | 59
Percentage of participants | 59.3 | 74.6 | 15.3

17. Secondary Outcome: Percentages of Participants Achieving a DLQI Score of 0 or 1 Over Time up to Week 52 - (Maintenance)
Description: as for outcome 16
Time Frame: Week 52
Population: Full Analysis Set (FAS) - All patients to whom study treatment was assigned.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg | Placebo
Number analyzed (Participants) | 59 | 60 | 28 | 28 | 3
Percentage of participants | 66.1 | 70.0 | 57.1 | 85.7 | 0.0

18. Secondary Outcome: Percentages of Participants With PASI 50, PASI 75, PASI 90, PASI 100 and IGA Mod 2011 0 or 1 Response After Week 52 (Observed Data)
Description: as for outcome 6
Time Frame: Week 160
Population: as for outcome 7
Measure: Number; unit: Percentages of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg
Number analyzed (Participants) | 61 | 60 | 28 | 28
Percentages of participants
  IGA 0/1 Week 160: number analyzed (Participants) | 16 | 24 | 10 | 15
  IGA 0/1 Week 160 | 43.8 | 58.3 | 20.0 | 73.3
  PASI 75 Week 160: number analyzed (Participants) | 16 | 24 | 10 | 15
  PASI 75 Week 160 | 93.8 | 87.5 | 70.0 | 86.7
  PASI 50 Week 160: number analyzed (Participants) | 16 | 24 | 10 | 15
  PASI 50 Week 160 | 100.0 | 100.0 | 70.0 | 100.0
  PASI 90 Week 160: number analyzed (Participants) | 16 | 24 | 10 | 15
  PASI 90 Week 160 | 62.5 | 70.8 | 40.0 | 73.3
  PASI 100 (n=16, 24, 10, 15) Week 160: number analyzed (Participants) | 16 | 24 | 10 | 15
  PASI 100 (n=16, 24, 10, 15) Week 160 | 31.3 | 45.8 | 20.0 | 60.0

19. Secondary Outcome: Absolute Change From Baseline for PASI Score After Week 52 (Observed Data)
Description: as for outcome 8
Time Frame: Week 160
Population: Full analysis set (FAS).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg
Number analyzed (Participants) | 61 | 60 | 28 | 28
Units on a scale | -18.7 (5.66) | -15.9 (4.58) | -12.7 (8.08) | -18.1 (5.49)

20. Secondary Outcome: Percentages of Participants in Each IGA Mod 2011 Category After Week 52 (Observed Data)
Description: as for outcome 10
Time Frame: Week 160
Population: Full analysis set (FAS).
Measure: Number; unit: Percentages of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg
Number analyzed (Participants) | 61 | 60 | 28 | 28
Percentages of participants
  clear Week 160: number analyzed (Participants) | 16 | 24 | 10 | 15
  clear Week 160 | 25.0 | 45.8 | 20.0 | 60.0
  almost clear Week 160: number analyzed (Participants) | 16 | 24 | 10 | 15
  almost clear Week 160 | 18.8 | 12.5 | 0.0 | 13.3
  mild Week 160: number analyzed (Participants) | 16 | 24 | 10 | 15
  mild Week 160 | 31.3 | 20.8 | 50.0 | 6.7
  moderate Week 160: number analyzed (Participants) | 16 | 24 | 10 | 15
  moderate Week 160 | 25.0 | 16.7 | 20.0 | 13.3
  severe Week 160: number analyzed (Participants) | 16 | 24 | 10 | 15
  severe Week 160 | 0.0 | 4.2 | 10.0 | 6.7

21. Secondary Outcome: Number of Participants Developing Treatment-emergent Anti-secukinumab Antibodies
Description: The development of anti-secunimubab anti-bodies decreases a participant's ability to respond to secukinumab treatment. The number of participants developing anti-secukinumab anti-bodies was measured from Baseline to week 216.
Time Frame: Baseline and at Week 12, 24, 52, 100, 148, 196, 208, and 216
Population: FAS
Measure: Number; unit: Number of participants
Groups:
- Placebo-AIN457 150 mg: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12, were re randomized to AIN457 150 mg for the remainder of the study.
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo-AIN457 150 mg | Placebo - AIN457 300mg | Placebo
Number analyzed (Participants) | 59 | 60 | 28 | 28 | 3
Number of participants | 1 | 2 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Treatment until Last Patient Last Visit, approximately 4 years.
Groups:
- Induction AIN457 150 mg: Patients received one secukinumab 150 mg s.c. injection plus one placebo secukinumab s.c. injection at each dosing. In the open label phase only one 150 mg s.c. injection at each dosing.
- Induction AIN457 300 mg: Patients received two secukinumab 150 mg s.c. injections at each dosing. In the open label phase only two 150 mg s.c. injections at each dosing.
- Induction Placebo; Entire Placebo: placebo secukinumab (2 s.c. injections) at each dosing
- Entire Any AIN457 150 mg: Includes all patients in the AIN457 150 mg and in the placebo- AIN457 150 mg treatment groups.
- Entire Any AIN457 300 mg: Includes all patients in the AIN457 300 mg and in the placebo- AIN457 300 mg treatment groups.
Arm/Group | Induction AIN457 150 mg | Induction AIN457 300 mg | Induction Placebo | Entire Any AIN457 150 mg | Entire Any AIN457 300 mg | Entire Placebo
Serious Adverse Events (participants affected / at risk) | 3/61 | 1/60 | 1/61 | 18/89 | 16/88 | 1/61
Other Adverse Events (participants affected / at risk) | 35/61 | 37/60 | 30/61 | 81/89 | 81/88 | 31/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction AIN457 150 mg (N=61) | Induction AIN457 300 mg (N=60) | Induction Placebo (N=61) | Entire Any AIN457 150 mg (N=89) | Entire Any AIN457 300 mg (N=88) | Entire Placebo (N=61)
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
ANGINA UNSTABLE (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
AORTIC VALVE STENOSIS (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
PALPITATIONS (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
POSTINFARCTION ANGINA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
AMAUROSIS FUGAX (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
CATARACT (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0
ASCITES (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
RECTAL PROLAPSE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
CHRONIC TONSILLITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
ERYSIPELAS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
MYELITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
BONE CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
DISLOCATION OF VERTEBRA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
HEART RATE IRREGULAR (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
ANOGENITAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
CAROTID ARTERY ANEURYSM (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
BLADDER PROLAPSE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
TRANSIENT ACANTHOLYTIC DERMATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction AIN457 150 mg (N=61) | Induction AIN457 300 mg (N=60) | Induction Placebo (N=61) | Entire Any AIN457 150 mg (N=89) | Entire Any AIN457 300 mg (N=88) | Entire Placebo (N=61)
EOSINOPHILIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 2 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 1 | 3 | 0
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 0 | 0 | 0 | 2 | 1 | 0
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 | 0 | 0 | 0 | 4 | 0
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 | 0 | 1 | 1 | 3 | 1
SINUS BRADYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 2 | 0 | 0
BLEPHARITIS (Eye disorders) | 0 | 2 | 0 | 0 | 4 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
DENTAL CARIES (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 0 | 6 | 7 | 0
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 3 | 0
TOOTHACHE (Gastrointestinal disorders) | 1 | 2 | 2 | 5 | 5 | 2
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 3 | 0
CYST (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
FATIGUE (General disorders) | 1 | 0 | 1 | 4 | 3 | 1
INJECTION SITE BRUISING (General disorders) | 0 | 1 | 0 | 1 | 4 | 0
INJECTION SITE HAEMATOMA (General disorders) | 0 | 0 | 2 | 1 | 3 | 2
INJECTION SITE PAIN (General disorders) | 0 | 1 | 0 | 1 | 2 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1 | 0 | 3 | 1 | 0
PYREXIA (General disorders) | 0 | 1 | 0 | 0 | 5 | 0
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 3 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 2 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 2 | 6 | 11 | 2
CANDIDA INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
CONJUNCTIVITIS (Infections and infestations) | 1 | 1 | 0 | 4 | 6 | 0
CYSTITIS (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
EAR INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 0
FOLLICULITIS (Infections and infestations) | 1 | 0 | 1 | 4 | 0 | 1
FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 1 | 2 | 6 | 7 | 2
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 3 | 2 | 0
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 0
HORDEOLUM (Infections and infestations) | 1 | 0 | 1 | 1 | 2 | 1
INFLUENZA (Infections and infestations) | 1 | 0 | 2 | 8 | 0 | 2
NASOPHARYNGITIS (Infections and infestations) | 14 | 19 | 9 | 37 | 39 | 9
ORAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 1 | 0 | 4 | 1
ORAL HERPES (Infections and infestations) | 1 | 0 | 0 | 4 | 4 | 0
OTITIS EXTERNA (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
PERIODONTITIS (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 0
PHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 5 | 5 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
PULPITIS DENTAL (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 0
PYURIA (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
RHINITIS (Infections and infestations) | 2 | 0 | 0 | 6 | 1 | 0
SINUSITIS (Infections and infestations) | 1 | 3 | 0 | 5 | 7 | 0
TINEA PEDIS (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0
TONSILLITIS (Infections and infestations) | 1 | 1 | 0 | 2 | 4 | 0
TOOTH ABSCESS (Infections and infestations) | 1 | 0 | 1 | 2 | 1 | 1
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 3 | 3 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1 | 17 | 9 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 2 | 3 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 3 | 2 | 0
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 1 | 0 | 0 | 4 | 1 | 0
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 4 | 0
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 4 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 3 | 0
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 2 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0
SUNBURN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 2 | 0
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 3 | 2 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 2 | 2 | 0
BLOOD URINE PRESENT (Investigations) | 0 | 0 | 0 | 0 | 3 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 2 | 0
LIVER FUNCTION TEST INCREASED (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
WEIGHT DECREASED (Investigations) | 0 | 0 | 1 | 2 | 0 | 1
WEIGHT INCREASED (Investigations) | 1 | 0 | 0 | 2 | 1 | 0
GOUT (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1 | 0
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 2 | 0
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 11 | 9 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 5 | 9 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 0
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 2 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3 | 4 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 3 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 3 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 3 | 1
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3 | 0 | 0
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 1 | 0
HEADACHE (Nervous system disorders) | 5 | 3 | 3 | 13 | 14 | 3
HYPOAESTHESIA (Nervous system disorders) | 0 | 1 | 0 | 2 | 1 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 0
ADJUSTMENT DISORDER WITH DEPRESSED MOOD (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 0
INSOMNIA (Psychiatric disorders) | 1 | 1 | 0 | 2 | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 6 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 1 | 0 | 0 | 2 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 5 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 5 | 10 | 2
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 3 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 4 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 4 | 8 | 2
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 5 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5 | 2 | 0
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
INTERTRIGO (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3 | 0 | 0
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 1
PITYRIASIS ROSEA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 4 | 2 | 3 | 7 | 2
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 6 | 7 | 1
SEBORRHOEA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 3 | 2 | 0
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2 | 0
HAEMATOMA (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 0
HYPERTENSION (Vascular disorders) | 3 | 1 | 4 | 4 | 10 | 4

LIMITATIONS AND CAVEATS:
Efficacy results after Wk 160 can't be interpreted meaningfully due to low # of evaluable patients. As per protocol, availability of AIN457 in participating countries led to discontinuation of most patients before they reached the later visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.